CLINICAL TRIAL: NCT04776044
Title: RESPIRE - A Randomized, Double-Blind, Placebo-Controlled, Multi-Centre Clinical Trial to Evaluate the Safety and Efficacy of ATR-002 in Adult Hospitalized Patients With COVID-19
Brief Title: Clinical Trial to Evaluate the Safety and Efficacy of ATR-002 in Adult Hospitalized Patients With COVID-19
Acronym: RESPIRE
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: general circumstances around COVID-19 and current availability of hospitalized patients
Sponsor: Atriva Therapeutics GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ATR-002-202
Record Dates: First submitted 2021-02-26; First posted 2021-03-01 (Actual); Last update posted 2022-09-22 (Actual); Status verified 2022-09

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — 2-(2-chloro-4-iodophenylamino)-N-3,4-difluorobenzoic acid

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo-controlled, multi-centre
Who Masked: Participant, Investigator
Masking Description: matching placebo tablets
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ATR-002 (Experimental): Participants will receive 900mg ATR-002 on day 1 (6 tablets with 150mg ATR-002; once daily), and 600mg ATR-002 on days 2 - 6 (4 tablets; once daily)
  Interventions: Drug: ATR-002
- Placebo (Placebo Comparator): Participants will receive matching tablets placebo on day 1 (6 tablets, once daily), and matching tablets placebo on days 2 - 6 (4 tablets per day, once daily)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ATR-002 — 150mg tablets for oral intake
  Arms: ATR-002
Drug: Placebo — matching tablets for oral intake
  Arms: Placebo

SUMMARY:
The purpose of the study is to assess the safety and efficacy of ATR-002 (in addition to standard-of-care) for the treatment of COVID-19

DETAILED DESCRIPTION:
After being informed about the study and potential risks, all patients giving written informed consent will be undergoing a 1-day screening to determine eligibility for study entry. At day 1, patients who meet the eligibility requirements will be randomized in a double-blind manner (participant and investigator) in a 1:1 ratio to ATR-002 (900mg day 1, 600mg days 2 - 6) or placebo (once daily)

ELIGIBILITY:
Inclusion Criteria:

1. Capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.
2. Study participant must be at least 18 years of age at the time of signing the ICF
3. Study participants with a laboratory confirmed diagnosis of SARS-CoV-2 infection presenting as moderate -to-severe COVID-19 requiring hospitalization for COVID-19 (Clinical Severity Status [3] or [4]) and for medical reasons (see Section 8). Patients presenting to the hospital without a laboratory confirmed SARS-CoV-2 infection will be tested locally for SARS-CoV-2 during the screening period. For sites in the EU: A CE certified SARS-CoV-2 PCR test kit is required to confirm infection. For sites outside the EU: SARS-CoV-2 PCR test kits certified according to local regulations are required to confirm infection.
4. Body weight at least 50 kg and a body mass index (BMI) ≥ 18.0 kg/m2 and < 40.0 kg/m2
5. Male or female Contraceptive use by women and men should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.
6. A female study participant is eligible to participate if she is not pregnant or breastfeeding, and one of the following conditions applies:

   1. She is not a WOCBP
   2. Is a WOCBP and is using a contraceptive method that is highly effective, with a failure rate of <1%, during the IMP period and for at least 4 weeks after the last dose of IMP. The investigator should evaluate the potential for contraceptive method failure (e.g., noncompliance, recently initiated) in relationship to the first dose of IMP.
7. A WOCBP must have a negative urine pregnancy test within 24 hours before the first dose of IMP.

   1. If a urine pregnancy test cannot be confirmed as negative (e.g., an ambiguous result), a serum pregnancy test is required locally. In such cases, the participant must not be randomized if the serum pregnancy result is positive.
   2. If a serum pregnancy test is required as per local regulations, a serum pregnancy test is required locally. In such cases, the participant must not be randomized if the serum pregnancy result is positive.
   3. The investigator is responsible for review of medical history, menstrual history, and recent sexual activity to decrease the risk for inclusion of a woman with an early undetectable pregnancy.
8. A male study participant is eligible to participate if:

   1. He is azoospermic
   2. The partner is not a WOCBP.
   3. The partner is a WOCBP and is using a contraceptive method that is highly effective, with a failure rate of <1%, during the IMP period and for at least 90 days after the last dose of IMP. The investigator should evaluate the potential for contraceptive method failure (e.g., noncompliance, recently initiated) in relationship to the first dose of IMP.
   4. He acknowledges that sperm donation is prohibited from the first dose of IMP until at least 90 days after the last dose of IMP.

Exclusion Criteria:

1. Patient's clinical condition is worsening rapidly.
2. Requiring ICU admission or ventilator support at screening or at randomization.
3. Suspected bacterial, fungal, viral, or other infection (besides COVID-19).
4. History of any of the following: malignant disease, autoimmune disease, or severe liver, kidney, blood, cardiac, pulmonary, neurological, or endocrine disease as judged by the investigator.
5. History of hypertension should have hypertension adequately controlled (BP < 140/90 mmHg) with appropriate anti-hypertensive treatment.
6. Clinically significant cardiac conduction abnormalities, including QTc prolongation of > 450 milliseconds
7. Family history of Long QT Syndrome.
8. Heart failure class 3, or 4, as defined by the New York Heart Association (NYHA).
9. History of acute coronary syndrome (including myocardial infarction), coronary angioplasty, or stenting within 24 weeks prior to screening.
10. Patients with implanted defibrillators or permanent pacemakers.
11. Poorly controlled diabetes mellitus with an HbA1c > 7.5 %.
12. Renal disease including glomerulonephritis, nephritic syndrome, Fanconi Syndrome, or renal tubular acidosis.
13. Renal failure requiring renal replacement therapy or moderate renal impairment as defined by having an estimated glomerular filtration rate (eGFR, CKD-EPI) < 45 ml/min/1.73m2.
14. Chronic Obstructive Pulmonary Disease (COPD) GOLD C, or D, or hospitalization for exacerbation of COPD within 24 weeks prior to screening.
15. Other chronic lung diseases including cystic fibrosis, neuromuscular diseases, severe chest wall deformities, interstitial lung diseases, outpatient chronic non-invasive ventilation due to chronic respiratory failure.
16. Asthma with a symptom control level of "uncontrolled", according to current GINA guidelines.
17. Currently suffering from diseases that seriously affect the immune system, such as: human immunodeficiency virus (HIV) infection, or the blood system, or splenectomy, or organ/ stem cell transplantation.
18. Known Hepatitis B or C infection.
19. Any medical condition, physical examination finding or laboratory abnormality that, in the opinion of the investigator, might confound the results of the study or pose an additional risk to the patient.
20. Alanine transaminase (ALT) or aspartate transaminase (AST) >3.0 x ULN.
21. Total bilirubin >1.0 x ULN (≥1.5 x ULN total bilirubin if known Gilbert's syndrome).
22. Taking concomitant medication metabolized by CYP2C8 and/ or CYP2C9.
23. Taking concomitant medication of any experimental treatment or use of marketed medications including off-label use, that are intended as specific treatment for COVID-19. Any such treatments must be washed out for 30 days or at least 5 half-lives prior to randomization, whichever is longer, unless a formal written standard of care policy document requires otherwise. Inclusion needs to be approved by the investigator and medical monitor.
24. Taking medication that may seriously affect the immune system, e.g., chemotherapy, unless considered and documented as standard of care (e.g., corticosteroids) to treat COVID-19.
25. Currently participating in other clinical trials or previous treatment with an investigational medicinal product within 5 half-lives or 30 days (whichever is longer) prior to randomization.
26. Known allergy or hypersensitivity to the IMP (including excipients).
27. Study participant is pregnant or breastfeeding.
28. Patient has been committed to an institution by virtue of an order issued either by the judicial or the administrative authorities.
29. Patient is an employee of the sponsor, or an employee of any third-party organization involved into the clinical trial, or an employee of the clinical trial site, or is dependent on the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 133 (Actual)
Dates: Start 2021-04-12 (Actual); Primary Completion 2022-06-06 (Actual); Study Completion 2022-08-09 (Actual)

PRIMARY OUTCOMES:
Clinical severity status on a 7-point ordinal scale | 15 days
  1. Not hospitalized, no limitations of activities
  2. Not hospitalized, limitations of activities
  3. Hospitalized, not requiring supplemental oxygen
  4. Hospitalized, requiring supplemental oxygen
  5. Hospitalized, on non-invasive ventilation or high flow oxygen devices
  6. Hospitalized, on invasive mechanical ventilation or ECMO
  7. Death

SECONDARY OUTCOMES:
Time from randomization to discharge from hospital | 90 days
Time to discharge from hospital or to score of ≤2 maintained for 24 hours in NEWS2, whichever occurs first | 90 days
Time to resolution of fever, defined as ≤36.6°C (axilla), ≤37.2°C (oral) or ≤37.8°C (rectal or tympanic) for at least 24 hours without antipyretics for 24 hours | 90 days
Time to SpO2 >94% on room air maintained for 24 hours | 90 days
Clinical severity status over the hospital period calculated as AUC from the 7-point ordinal scale at Days 3, 5, 8, 11, 15 and 30 | at days 3, 5, 8, 11 and 30

CONTACTS AND LOCATIONS:
Overall Officials: University Clinic Frankfurt M Medical Clinic, Principal Investigator — Centre of Pneumology
Locations (40):
- Germany (10):
  - Atriva study site 49006, Augsburg
  - Atriva study site 49001, Berlin
  - Atriva study site 49013, Berlin
  - Atriva study site 49011, Dresden
  - Atriva study site 49003, Frankfurt
  - Atriva study site 49008, Frankfurt
  - Atriva study site 49009, Freiburg im Breisgau
  - Atriva study site 49007, Halle
  - Atriva study site 49004, Münster
  - Atriva study site 49012, Rostock
- India (7):
  - Atriva study site 91002, Ahmedabad
  - Atriva study site 91001, Aligarh
  - Atriva study site 91011, Aurangabad
  - Atriva study site 91008, Mumbai
  - Atriva study site 91009, Mumbai
  - Atriva study site 91003, New Delhi
  - Atriva study site 91004, Raipur
- Netherlands (2):
  - Atriva study site 31001, Eindhoven
  - Atriva study site 31002, Tilburg
- Poland (3):
  - Atriva study site 48002, Bolesławiec
  - Atriva study site 48004, Bolesławiec
  - Atriva study site 48003, Warsaw
- Romania (5):
  - Atriva study site 40006, Bucharest
  - Atriva study site 40002, Iași
  - Atriva study site 40004, Sibiu
  - Atriva study site 40008, Suceava
  - Atriva study site 40003, Timișoara
- South Africa (6):
  - Atriva study site 27005, Benoni
  - Atriva study site 27002, Cape Town
  - Atriva study site 27003, George
  - Atriva study site 27006, KwaZulu
  - Atriva study site 27007, Mayville
  - Atriva study site 27008, Pretoria
- Spain (7):
  - Atriva study site 34001, Barcelona
  - Atriva study site 34011, Lleida
  - Atriva study site 34002, Madrid
  - Atriva study site 34005, Madrid
  - Atriva study site 34008, Madrid
  - Atriva study site 34010, Pontevedra
  - Atriva study site 34004, Valencia

REFERENCES:
- [Derived] Rohde G, Stenglein S, Prozesky H, Manudhane G, Sandulescu O, Bauer M, Overend T, Koch W, Neuschwander D, Planz O, Torres A, Witzenrath M. Efficacy and safety of zapnometinib in hospitalised adult patients with COVID-19 (RESPIRE): a randomised, double-blind, placebo-controlled, multicentre, proof-of-concept, phase 2 trial. EClinicalMedicine. 2023 Oct 4;65:102237. doi: 10.1016/j.eclinm.2023.102237. eCollection 2023 Nov. PMID 38106555